CLINICAL TRIAL: NCT02926638
Title: A Phase II/III Randomized Study of Rilotumumab Plus Erlotinib Versus Erlotinib as Second Line Therapy for C-Met Positive Patients With Stage IV Squamous Cell Lung Cancer (Lung-Map Sub-Study)
Brief Title: Lung-MAP: Rilotumumab and Erlotinib Hydrochloride or Erlotinib Hydrochloride Alone as Second-Line Therapy in Treating Patients With Recurrent Stage IV Squamous Cell Lung Cancer and Positive Biomarker Matches
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Drug company decided to terminate all sponsored clinical studies involving rilotumumab.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1400E; NCI-2014-01382 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1400E; S1400E (Other: SWOG); S1400E (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2016-05-06; First posted 2016-10-06 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: MET Positive; Recurrent Squamous Cell Lung Carcinoma; Stage IV Squamous Cell Lung Carcinoma AJCC v7
MeSH Terms: interventions — Erlotinib Hydrochloride; rilotumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Arm I (rilotumumab, erlotinib) (Experimental): Patients receive rilotumumab IV over 60-120 minutes on day 1 and erlotinib hydrochloride PO daily. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. (CLOSED TO ACCRUAL AND INTERVENTION 11/25/2014)
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis; Biological: Rilotumumab
- Arm II (erlotinib) (Active Comparator): Patients receive erlotinib hydrochloride PO daily. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. (CLOSED TO ACCRUAL AND INTERVENTION 11/25/2014)
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Rilotumumab — Given IV
  Other Names: AMG 102; Anti-HGF Monoclonal Antibody AMG 102; Fully Human Anti-HGF Monoclonal Antibody AMG 102
  Arms: Arm I (rilotumumab, erlotinib)

SUMMARY:
This randomized phase II/III compares rilotumumab when given together with erlotinib hydrochloride against erlotinib hydrochloride alone in treating patients with stage IV squamous cell lung cancer that has come back after previous treatment. This is a sub-study that includes all screened patients positive for the met proto-oncogene (MET)/hepatocyte growth factor (HGF) biomarker. HGF can interact with MET and can cause tumor cells to grow more quickly. Rilotumumab may decrease the activity of HGF and may be able to shrink tumors. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving rilotumumab with erlotinib hydrochloride works better than erlotinib hydrochloride alone (standard treatment) in treating squamous cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if there is sufficient evidence to continue to the phase III component of S1400E by comparing investigator-assessed progression-free survival (IA-PFS) between rilotumumab plus erlotinib versus erlotinib in patients registered to S1400E. (Phase II) II. To determine if there is both a statistically and clinically-meaningful difference in IA-PFS between patients randomized to receive rilotumumab plus erlotinib versus erlotinib. (Phase III) III. To compare overall survival (OS) in patients randomized to rilotumumab plus erlotinib versus erlotinib. (Phase III)

SECONDARY OBJECTIVES:

I. To compare response rates (confirmed and unconfirmed, complete and partial responses) among patients randomized to receive rilotumumab plus erlotinib versus erlotinib. (Phase II) II. To evaluate the frequency and severity of toxicities associated with rilotumumab plus erlotinib versus erlotinib. (Phase II) III. To compare the response rates (confirmed and unconfirmed, complete and partial) among patients randomized to receive rilotumumab plus erlotinib versus erlotinib. (Phase III) IV. To evaluate the frequency and severity of toxicities associated with rilotumumab plus erlotinib versus erlotinib. (Phase III)

TERTIARY OBJECTIVES:

I. To evaluate the treatment arm randomization acceptance rate within each treatment arm of S1400E defined as the percentage of patients randomized to a treatment arm that receive any protocol treatment.

II. To identify additional predictive or prognostic tumor/blood biomarkers beyond the chosen biomarker.

III. To identify potential resistance biomarkers at disease progression. IV. To establish a tissue/blood repository from patients with refractory squamous cell cancer.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (CLOSED TO ACCRUAL AND INTERVENTION11/25/2014): Patients receive rilotumumab intravenously (IV) over 60-120 minutes on day 1 and erlotinib hydrochloride orally (PO) daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II (CLOSED TO ACCRUAL AND INTERVENTION11/25/2014): Patients receive erlotinib hydrochloride PO daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, all patients will be followed until death or 3 years after sub-study registration, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all SCREENING/PRE-SCREENING and SUB-STUDY REGISTRATION COMMON ELIGIBILITY CRITERIA as specified in S1400: Phase II/III Biomarker-Driven Master Protocol for Previously Treated Squamous Cell Lung Cancer (Lung-Map)
* Patients must be assigned to S1400E; S1400E biomarker eligibility defined as C-MET positive is defined as follows:

  * Analyte: C-MET
  * Assay: Immunohistochemistry (IHC)
  * Eligible definition: IHC positive based on Dako MET-IHC pharm DX kit
* If randomized to arm I rilotumumab plus erlotinib, patients must be willing to provide blood specimens for anti-rilotumumab anti-body testing
* Patients must not have peripheral edema > grade 1 at the time of sub-study registration
* Patients must not have received prior treatment with MET pathway, inhibitors or EGFR inhibitors (e.g., erlotinib)
* Patients must have total bilirubin =< 1.5 x institutional upper limits of normal (IULN) within 28 days prior to sub-study registration
* Patients must not have abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjorgren?s syndrome), congenital abnormality (e.g., Fuch?s dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal-Rose), and/or abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Patients must not be taking, nor plan to take while on protocol treatment and for 14 days post the last dose of study treatment, drugs, herbal supplements or foods that are known to be strong/moderate CYP3A4 substrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2015-01-12 (Actual); Study Completion 2016-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki Papadimitrakopoulou, Principal Investigator — SWOG Cancer Research Network
Locations (627):
- United States (627):
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Kaiser Permanente, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Feather River Cancer Center, Paradise, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Medical Oncology and Hematology Group PC-Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale-New Haven Hospital Saint Raphael Campus, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Charlotte Hungerford Hospital Center for Cancer Care, Torrington, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Florida Health Science Center ?? Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Leeward, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Hematology Oncology Consultants Limited, Naperville, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - IU Health Central Indiana Cancer Centers-Fishers, Fishers, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - LSU Healthcare Network/Saint Charles, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Mercy Hospital, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - York Hospital, York Village, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Cancer Center-Golden Triangle, Columbus, Mississippi
  - Boston Baskin Cancer Center-Grenada, Grenada, Mississippi
  - Family Cancer Center-Oxford, Oxford, Mississippi
  - Family Cancer Center-Southhaven, Southaven, Mississippi
  - Baptist Memorial Hospital-Desoto, Southhaven, Mississippi
  - Baptist Cancer Institute-Starkville, Starkville, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Faith Regional Medical Offices West, Norfolk, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Oncology Hematology West, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Regional West Medical Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Alpine Hematology-Oncology, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Reno Oncology Consultants, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - PinnacleHealth Cancer Center-Community Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-St. Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Georgetown Hospital System, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Boston Baskin Cancer Center-Bartlett, Bartlett, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology Associates PC, Winchester, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology SC-Appleton, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated early and thus no manuscript will be forthcoming. Outcomes were not analyzed.
Period: Overall Study
Arm/Group | Arm I (Rilotumumab, Erlotinib) | Arm II (Erlotinib)
Started | 4 | 5
Eligible | 3 | 5
Completed | 0 | 0
Not Completed | 4 | 5
Not completed — Progression | 2 | 5
Not completed — Ineligible | 1 | 0
Not completed — Not protocol specified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Rilotumumab, Erlotinib) | Arm II (Erlotinib) | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Median (Full Range); unit: years] | 73 [69.3 to 75.8] | 71.6 [48.7 to 79.5] | 72.3 [48.7 to 79.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Investigator-assessed Progression-free Survival Between Arms
Description: A stratified (using randomization stratification factors) log-rank test will be used to test the primary hypotheses related to investigator-assessed progression-free survival, comparing the two treatment arms.
Time Frame: From date of sub-study registration to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause, assessed up to 18 months since completion of accrual
Population: This study was terminated early and thus no manuscript is forthcoming. Outcomes were not analyzed.
Arm/Group | Arm I (Rilotumumab, Erlotinib) | Arm II (Erlotinib)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Objective Response Rate (Confirmed and Unconfirmed, Complete and Partial) Between Arms
Time Frame: Up to 3 years
Population: This study was terminated early and thus no manuscript is forthcoming. Outcomes were not analyzed.
Arm/Group | Arm I (Rilotumumab, Erlotinib) | Arm II (Erlotinib)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Frequency and Severity of Toxicities Associated With Investigational Therapy Versus Standard of Care
Time Frame: Up to 3 years
Population: This study was terminated early and thus no manuscript is forthcoming. Outcomes were not analyzed.
Arm/Group | Arm I (Rilotumumab, Erlotinib) | Arm II (Erlotinib)
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Treatment Arm Randomization Acceptance Rate
Description: Monitored by the percentage of patients that receive at least one dose of the treatment they are randomized to.
Time Frame: Up to 3 years
Population: This study was terminated early and thus no manuscript is forthcoming. Outcomes were not analyzed.
Arm/Group | Arm I (Rilotumumab, Erlotinib) | Arm II (Erlotinib)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: This study was terminated early and thus no manuscript is forthcoming. Outcomes were not analyzed. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Arm I (Rilotumumab, Erlotinib) | Arm II (Erlotinib)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No